CLINICAL TRIAL: NCT00809445
Title: HIV Rapid Testing and Counseling in Drug Abuse Treatment Programs in the U.S.
Brief Title: Rapid HIV Testing and Counseling in Drug Abuse Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Daniel J Feaster, Associate Professor of Biostatistics, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20080379; U10DA013720 (NIH)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2014-09

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HIV rapid test & counseling (Experimental): Participants will be offered an oral fluid HIV rapid test (via oral swab) and brief prevention counseling that addresses both risk reduction and motivation to be HIV tested based on an evidence-based counseling approach (Project RESPECT-2 counseling). Prior to receiving testing, study participants must first provide consent for HIV testing. Consent for testing will be obtained through a second consent form required of all participants who wish to proceed with the HIV test.
  Interventions: Behavioral: On-site HIV rapid test and brief, prevention counseling
- HIV rapid test and info (Experimental): Participants will be offered an oral fluid HIV rapid test (via oral swab). Prior to receiving testing, study participants must first provide consent for HIV testing. Again, consent for testing will be obtained through a second consent form required of all participants who wish to proceed with the HIV test. Participants will receive rapid HIV testing and test results after signing the consent to be tested. In both Groups 1 and 2, participants who test reactive (preliminary positive) will be counseled on the sexual risk behaviors associated with transmission of HIV and the acquisition of STDs, as is current clinical practice with those testing HIV positive. Confirmed positives will be linked to HIV primary care.
  Interventions: Behavioral: On- site HIV rapid test & information
- HIV testing referral (Active Comparator): Participants randomized to group 3 will receive a referral list for HIV community-testing agencies. Each CTP site will have previously prepared an extensive referral list of testing sites in the surrounding geographic area. By virtue of their status as patients in the CTPs, they will receive whatever HIV testing and HIV education referrals the CTPs normally provide to their patients. This is the standard of care at CTPs that do not provide on-site testing.
  Interventions: Behavioral: Referral for off-site HIV testing

INTERVENTIONS:
Behavioral: On-site HIV rapid test and brief, prevention counseling — Participants will be offered an on-site oral fluid HIV rapid test with brief prevention counseling that addresses both risk reduction and motivation to be HIV tested based on an evidence-based counseling approach.
  Arms: HIV rapid test & counseling
Behavioral: On- site HIV rapid test & information — Participants will be offered an on-site oral fluid HIV rapid test with basic info.
  Arms: HIV rapid test and info
Behavioral: Referral for off-site HIV testing — Participants will be offered a referral list of HIV testing agencies in the community.
  Arms: HIV testing referral

SUMMARY:
This is a randomized controlled clinical trial in which adults receiving drug abuse treatment will be recruited to participate in a multi-center HIV testing and counseling study. The purpose of this study is to assess the relative effectiveness of three HIV testing strategies on increasing receipt of test results: (1) on-site HIV rapid testing with brief, participant-tailored prevention counseling, (2) on-site HIV rapid testing with information only, and (3) referral for off-site HIV testing. The study will also assess the effectiveness of the three testing strategies in reducing HIV risk behaviors.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial in which individuals receiving drug abuse treatment will be recruited to participate in a multi-center HIV testing and counseling study. The purpose of this study is to assess the relative effectiveness of three HIV testing strategies on increasing receipt of HIV test results: (1) on-site HIV rapid testing with brief, participant-tailored prevention counseling, (2) on-site HIV rapid testing with information only, and (3) referral for off-site HIV testing. The study will also assess the effectiveness of the three testing strategies in reducing HIV sexual risk behaviors. Injection drug risk behavior will be a secondary outcome. Participants will complete a baseline assessment to report their demographics, HIV testing history and sexual and drug-using risk behaviors, and will be randomized to one of three groups. At one month post-randomization, participants will complete a follow-up assessment to determine whether or not they received their HIV test results. At six months post-randomization, participants will complete a follow-up assessment to assess any changes in their HIV sexual risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* HIV-negative or HIV status unknown
* No receipt of results from HIV test initiated within last 12 months
* Be able to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1281 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Metsch, Ph.D., Principal Investigator — Columbia University; Grant Colfax, M.D., Principal Investigator — PATH
Locations (12):
- United States (12):
  - La Frontera Center, Inc., Tucson, Arizona
  - Midwestern Connecticut Council on Alcoholism, Danbury, Connecticut
  - Wheeler Clinic, Plainville, Connecticut
  - Glenwood Life Counseling Center, Baltimore, Maryland
  - Gibson Recover Centers, Cape Girardeau, Missouri
  - The Life Link, Santa Fe, New Mexico
  - Daymark Recovery Services, Inc., Salisbury, North Carolina
  - CODA, Portland, Oregon
  - Addiction Medicine Services (Western Psychiatric Institute), Pittsburgh, Pennsylvania
  - Morris Village Alcohol and Drug Treatment Center, Columbia, South Carolina
  - Lexington / Richland Alcohol and Drug Abuse Council, Columbia, South Carolina
  - Chesterfield CSB Substance Abuse Service, Chesterfield, Virginia

REFERENCES:
- [Result] Metsch LR, Feaster DJ, Gooden L, Matheson T, Mandler RN, Haynes L, Tross S, Kyle T, Gallup D, Kosinski AS, Douaihy A, Schackman BR, Das M, Lindblad R, Erickson S, Korthuis PT, Martino S, Sorensen JL, Szapocznik J, Walensky R, Branson B, Colfax GN. Implementing rapid HIV testing with or without risk-reduction counseling in drug treatment centers: results of a randomized trial. Am J Public Health. 2012 Jun;102(6):1160-7. doi: 10.2105/AJPH.2011.300460. Epub 2012 Apr 19. PMID 22515871
- [Result] Schackman BR, Metsch LR, Colfax GN, Leff JA, Wong A, Scott CA, Feaster DJ, Gooden L, Matheson T, Haynes LF, Paltiel AD, Walensky RP. The cost-effectiveness of rapid HIV testing in substance abuse treatment: results of a randomized trial. Drug Alcohol Depend. 2013 Feb 1;128(1-2):90-7. doi: 10.1016/j.drugalcdep.2012.08.009. Epub 2012 Sep 9. PMID 22971593
- [Derived] Schackman BR, Leff JA, Barter DM, DiLorenzo MA, Feaster DJ, Metsch LR, Freedberg KA, Linas BP. Cost-effectiveness of rapid hepatitis C virus (HCV) testing and simultaneous rapid HCV and HIV testing in substance abuse treatment programs. Addiction. 2015 Jan;110(1):129-43. doi: 10.1111/add.12754. PMID 25291977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults receiving drug abuse treatment in drug treatment clinics were recruited, screened for eligibility, and randomized from Jan - May 2009 into 1 of 3 arms: 1) on-site HIV rapid testing with counseling; 2) on-site HIV rapid testing with information only; and 3) referral for off-site HIV testing. Participants were then followed at 1 and 6 months.
Pre-assignment Details: 2473 patients were assessed for eligibility. Of these, 1313 were eligible and 1281 were randomized; 32 screened eligible, but were not randomized due to: failure to return to the study (n=30), lying about HIV status (n=1) and completing the baseline after the enrollment period closed (n=1).
Groups:
- HIV Testing Referral: Referral for off-site HIV testing : Participants will be offered a referral list of HIV testing agencies in the community.
- HIV Rapid Test & Counseling: On-site HIV rapid test and brief, prevention counseling : Participants will be offered an on-site oral fluid HIV rapid test with brief prevention counseling that addresses both risk reduction and motivation to be HIV tested based on an evidence-based counseling approach.
- HIV Rapid Test and Info: On- site HIV rapid test & information : Participants will be offered an on-site oral fluid HIV rapid test with basic info.
Period: 1 Month Follow-up
Arm/Group | HIV Testing Referral | HIV Rapid Test & Counseling | HIV Rapid Test and Info
Started | 429 | 433 | 419
Completed | 427 | 429 | 415
Not Completed | 2 | 4 | 4
Not completed — Lost contact | 1 | 2 | 1
Not completed — Withdrew consent | 1 | 1 | 1
Not completed — Death | 0 | 1 | 1
Not completed — Incarcerated | 0 | 0 | 1
Period: 6 Month Follow-up
Arm/Group | HIV Testing Referral | HIV Rapid Test & Counseling | HIV Rapid Test and Info
Started | 429 | 433 | 419
Completed | 405 | 410 | 395
Not Completed | 24 | 23 | 24
Not completed — Lost contact | 16 | 14 | 14
Not completed — Death | 2 | 1 | 1
Not completed — Incarcerated | 6 | 8 | 8
Not completed — Withdrew consent | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants were recruited from 12 community-based drug treatment programs. The Baseline Analysis Population represents the 1281 participants who completed baseline and were subsequently randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Testing Referral | HIV Rapid Test & Counseling | HIV Rapid Test and Info | Total
Number analyzed (Participants) | 429 | 433 | 419 | 1281
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1 | 2
  Between 18 and 65 years | 425 | 429 | 415 | 1269
  >=65 years | 3 | 4 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.81 (10.76) | 39.62 (11.19) | 39.56 (11.77) | 40.00 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 170 | 160 | 503
  Male | 256 | 263 | 259 | 778
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 89 | 88 | 86 | 263
  White | 278 | 277 | 271 | 826
  American Indian/Alaskan Native | 9 | 13 | 11 | 33
  Mixed race | 34 | 34 | 30 | 98
  Other | 19 | 21 | 21 | 61
  Hispanic | 51 | 49 | 47 | 147
Region of Enrollment [Number; unit: participants]
  United States | 429 | 433 | 419 | 1281

OUTCOME MEASURES:

1. Primary Outcome: Self-Report Receipt of HIV Test Results
Description: The HIV testing primary outcome is self-reported receipt of HIV test results. This will be measured at one month post-randomization for all participants. We recognize that there are three potential HIV testing behaviors that could be evaluated in this study: acceptance of HIV testing, completion of HIV testing, and receipt of HIV testing results. Acceptance of testing refers to whether or not a participant would accept the offer of an HIV test. Completion of testing refers to whether or not a participant completes the HIV test. Receipt of HIV test results refers to whether or not a participant self-reports having received the results of the HIV test.
Time Frame: One month post-randomization
Population: All randomized participants who provided self-report of either receipt or non-receipt of testing results at one month follow-up are included. Note that 3, 5, and 6 participants who completed a one-month follow-up did not provide this self-report in HIV testing referral, HIV rapid test and counseling, and HIV rapid test and info, respectively
Measure: Number; unit: participants
Arm/Group | HIV Testing Referral | HIV Rapid Test & Counseling | HIV Rapid Test and Info
Number analyzed (Participants) | 424 | 424 | 409
participants | 78 | 338 | 347
Statistical Analysis 1: Comparison: HIV Testing Referral vs HIV Rapid Test & Counseling vs HIV Rapid Test and Info; Hypothesis: The HIV rapid testing arms would have a higher rate of HIV testing than the HIV testing referral arm. Thus there is one comparison: HIV rapid test & counseling+HIV rapid test and info versus HIV testing referral; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — a-prior threshold for statistical significance is .025; Risk Ratio (RR) = 4.52, 97.5% CI 2-sided [3.57 to 5.72] — The numerator is the two HIV rapid testing arms The denominator is the HIV testing referral arm

2. Primary Outcome: Number of Risky Sexual Behaviors
Description: The sexual risk behavior primary outcome is self-reported sexual risk behavior, which will be measured at baseline and six months post-randomization as the self-reported number of unprotected sex acts (vaginal or anal sex without a condom).
Time Frame: Six months post-randomization
Population: All randomized participants who provided self-report of number of unprotected sex acts (vaginal or anal sex without a condom) at six-month follow-up are included.
Measure: Mean (Standard Deviation); unit: number of unprotected sex acts
Arm/Group | HIV Testing Referral | HIV Rapid Test & Counseling | HIV Rapid Test and Info
Number analyzed (Participants) | 387 | 385 | 371
number of unprotected sex acts | 20.5 (49.8) | 21.3 (47.6) | 21.3 (44.8)
Statistical Analysis 1: Comparison: HIV Testing Referral vs HIV Rapid Test & Counseling vs HIV Rapid Test and Info; Hypothesis: The HIV rapid testing arms would have a lower rate of unprotected sexual episodes than the HIV testing referral arm. Thus there is one comparison: HIV rapid test & counseling+HIV rapid test and info versus HIV testing referral; Test type: Superiority or Other; p = 0.39, generalized estimating equations (GEE) — a-priori threshold for statistical significance is .025; incidence rate raios (IRR) = 1.04, 97.5% CI 2-sided [0.95 to 1.14] — Numerator includes the two HIV rapid testing groups Denominator is the HIV testing referral group
Statistical Analysis 2: Comparison: HIV Rapid Test & Counseling vs HIV Rapid Test and Info; The data analysis information presented is for the comparison of the 2 on-site testing groups. Hypothesis: HIV rapid test and counseling group will have fewer unprotected sexual acts than will HIV rapid test and info group; Test type: Superiority or Other; p = 0.81, Generalized estimating equations (GEE) — a-priori threshold for statistical significance is .025; Incidence rate ratio (IRR) = 1.03, 97.5% CI 2-sided [0.84 to 1.26] — Numerator is the HIV rapid test and counseling arm Denominator is the HIV rapid test and info arm

3. Secondary Outcome: Sharing of Needles Used in Drug Use
Description: Change in sharing of needles. The number of individuals reporting needle sharing at baseline and 6-month follow-up were measured and the change in sharing of needles assessed.
Time Frame: Six months
Measure: Number; unit: n of people changing needle sharing
Arm/Group | HIV Testing Referral | HIV Rapid Test & Counseling | HIV Rapid Test and Info
Number analyzed (Participants) | 401 | 402 | 385
n of people changing needle sharing
  Number discontinuing sharing | 17 | 32 | 24
  Number initiating sharing | 2 | 1 | 6
Statistical Analysis 1: Comparison: HIV Testing Referral vs HIV Rapid Test & Counseling vs HIV Rapid Test and Info; Test type: Superiority or Other; p = 0.044, Chi-squared — a priori threshold for significance was .05; Note that this is a 3 by 3 chi-square: the 3 conditions by discontinued sharing needles /no change in sharing needles/initiated sharing needles

4. Secondary Outcome: Self-Report of Ever Having Been Tested
Description: The HIV testing secondary outcomes are all binary (Yes/No). The below data represents self-reported completion of HIV test by 1 month.
Time Frame: 1 month post-randomization
Population: Number reporting having taken an HIV test, whether they received results or not, at one month follow-up. Note that 3, 5, and 6 participants who completed a one-month follow-up did not provide this self-report in HIV testing referral, HIV rapid test and counseling, and HIV rapid test and info, respectively
Measure: Number; unit: participants
Arm/Group | HIV Testing Referral | HIV Rapid Test & Counseling | HIV Rapid Test and Info
Number analyzed (Participants) | 424 | 424 | 409
participants | 103 | 344 | 352
Statistical Analysis 1: Comparison: HIV Testing Referral vs HIV Rapid Test & Counseling vs HIV Rapid Test and Info; Test type: Superiority or Other; p < 0.0001, Chi-squared — a-priori threshold for statistical significance is .05; chi-square = 428.2466, Df=2

ADVERSE EVENTS:
Time Frame: AE will be reported within 7 days of the site becoming aware of the event. 24 hr expedited reporting is required for reportable serious adverse events. Lead investigators and the NIDA assigned Safety Monitor will be notified within 24 hours.
Description: Research staff will use a standard checklist to document adverse events at each research visit following randomization. This information will be collected and documented in the study database via CRF.
Arm/Group | HIV Testing Referral | HIV Rapid Test & Counseling | HIV Rapid Test and Info
Serious Adverse Events (participants affected / at risk) | 2/429 | 2/433 | 2/419
Other Adverse Events (participants affected / at risk) | 0/429 | 0/433 | 0/419
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV Testing Referral (N=429) | HIV Rapid Test & Counseling (N=433) | HIV Rapid Test and Info (N=419)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Overdose (General disorders) | 0 (0) | 0 (0) | 2 (2)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) — unknown cause; "general disorders" selected as default

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No